CLINICAL TRIAL: NCT00186394
Title: High Dose Chemotherapy and Allogeneic Hematopoietic Cell Transplantation for Non-Hodgkin's Lymphoma
Brief Title: High Dose Chemotherapy and Allogeneic Hematopoietic Cell Transplant for Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Wen-Kai Weng, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT4L; 76679; BMT4L; NCT00186394
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Lymphoma, Non-Hodgkin; Blood and Marrow Transplant (BMT); Lymphomas: Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Procedure: ablative allogeneic hematopoietic cell transplantation

SUMMARY:
To evaluate the role of allogeneic hematopoietic cell transplantation in the treatment of NHL.

DETAILED DESCRIPTION:
To determine safety and toxicity of a regimen of high dose chemotherapy with allogeneic peripheral blood progenitor cell transplantation; determine the efficacy of the procedure by following clinical outcomes and quality of life measures; and evaluate graft versus host disease incidence and severity with regimen.

ELIGIBILITY:
Inclusion Criteria:Morphologically confirmed relapsed non-Hodgkin's lymphoma

Age: >18 and <61 years of age

Signed informed consent Exclusion Criteria:Hepatic dysfunction defined by serum transaminases >2.5X normal values

Serum creatinine of > 2 mg/dl or creatinine clearance < 60 ml/min

Diseases other than non-Hodgkin's lymphoma

Prior bone marrow transplant procedure

Severe psychological or medical illness

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2000-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety
Toxicity
Efficacy

SECONDARY OUTCOMES:
Incidence of acute and chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kai Weng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States